CLINICAL TRIAL: NCT03137667
Title: Efficacy Study of School-located Influenza Vaccination Clinics to Increase Influenza Vaccination Rates in Monroe County, New York
Brief Title: School-located Influenza Vaccination Clinics for Adolescents
Acronym: SKIPP RCT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Rochester (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5R18HS021163-02 (AHRQ)
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Childhood Influenza Vaccination; School-located Influenza Vaccination
Keywords: Influenza Vaccination Rates

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator is not aware of the allocation at the level of the patient. In addition, the investigator is not involved in vaccine verification (data collection involving patient-level vaccination status)
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No school-located influenza vaccination clinic
- School-located Influenza Vaccination (Experimental): Children in intervention schools were offered a chance to receive influenza vaccination at a school-located influenza vaccination clinic, if their parent or legal guardian provided permission
  Interventions: Other: School-located Influenza Vaccination

INTERVENTIONS:
Other: School-located Influenza Vaccination — Children in the intervention arm are enrolled in schools in Monroe County, New York that are offering school-located influenza vaccination clinics during school hours
  Arms: School-located Influenza Vaccination

SUMMARY:
A cluster-randomized trial (clustering by school) was conducted in Monroe County, NY. Twenty middle and high schools were paired based on several characteristics and randomized within pairs to receiving a school-based influenza vaccination clinic or not (control).

DETAILED DESCRIPTION:
The overarching goal of the study was to evaluate the effectiveness and cost-effectiveness of offering school-based influenza vaccination clinics during school hours on influenza vaccination rates. A cluster-randomized trial (clustering by school) was conducted in Monroe County, NY. Twenty middle and high schools were paired based on several characteristics including urban/suburban,school grade-span (6-8th, 9-12th), school size, percent of students eligible for free or reduced school lunch, and influenza vaccination rates in the previous season among students in the school. School were randomized within pairs, with one school offering a school-based influenza vaccination clinic or and one school not offering the clinic (control).

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled students of a participating school

Exclusion Criteria:

* Not a currently enrolled student of a participating school

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17650 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Influenza vaccination status as recorded in the NY state registry (NYSIIS) | Within one year
  Vaccination status for the 2014/2015 influenza season will be assessed. The vaccination date will be recorded, as well as the provider name, to determine whether vaccine was received at the school-located influenza clinic

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yoo BK, Schaffer SJ, Humiston SG, Rand CM, Goldstein NPN, Albertin CS, Concannon C, Szilagyi PG. Cost effectiveness of school-located influenza vaccination programs for elementary and secondary school children. BMC Health Serv Res. 2019 Jun 24;19(1):407. doi: 10.1186/s12913-019-4228-5. PMID 31234842
- [Derived] Schaffer SJ, Rand CM, Humiston SG, Concannon C, Hightower AD, Albertin C, Szilagyi PG. Practical considerations in developing a successful school-located influenza vaccination (SLIV) program. Vaccine. 2019 Apr 10;37(16):2171-2173. doi: 10.1016/j.vaccine.2019.01.088. Epub 2019 Mar 13. No abstract available. PMID 30878250
- [Derived] Szilagyi PG, Schaffer S, Rand CM, Goldstein NPN, Younge M, Mendoza M, Albertin CS, Concannon C, Graupman E, Hightower AD, Yoo BK, Humiston SG. Text Message Reminders for Child Influenza Vaccination in the Setting of School-Located Influenza Vaccination: A Randomized Clinical Trial. Clin Pediatr (Phila). 2019 Apr;58(4):428-436. doi: 10.1177/0009922818821878. Epub 2019 Jan 2. PMID 30600690